CLINICAL TRIAL: NCT03742791
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Titration Study to Evaluate the Safety, Tolerability and Pharmacokinetics of TS-134 Administered Orally to Healthy Male and Female Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of 14-day Multiple Dose Titrations of TS-134 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical R&D Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TS134-US102
Record Dates: First submitted 2018-10-18; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
Keywords: TS-134, multiple dose, titration

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TS-134 (Experimental): Healthy adult subjects will be prospectively assigned to 1 of 6 cohorts. Within each cohort, 10 subjects per cohort will be randomized in a 4:1 ratio (8 active + 2 placebo) to receive daily doses of TS-134 or placebo for 14 days in a fed state, with ascending titrated dose levels ranging from 5 mg to 80 mg, depending on the assigned cohort. The maximum daily dose shall not exceed 80 mg.
  Interventions: Drug: TS-134
- Placebo (Placebo Comparator): Healthy adult subjects will be prospectively assigned to 1 of 6 cohorts. Within each cohort, 10 subjects per cohort will be randomized in a 4:1 ratio (8 active + 2 placebo) to receive daily doses of TS-134 or placebo for 14 days in a fed state, with ascending titrated dose levels ranging from 5 mg to 80 mg, depending on the assigned cohort. The maximum daily dose shall not exceed 80 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TS-134 — 5 mg to 80 mg oral solution
  Arms: TS-134
Drug: Placebo — Matched Placebo oral solution
  Arms: Placebo

SUMMARY:
This is a Phase 1 study involving multiple dose titrations of TS-134 in healthy male and female subjects. The safety, tolerability and pharmacokinetics of multiple dose titrations of TS-134 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female participants between 18 and 55 years of age
* Body weight greater than or equal to 45 kg
* Body Mass Index (BMI) greater than or equal to 18 and less than or equal to 30 kg/m^2

Exclusion Criteria:

* Female participants who are pregnant, intend to become pregnant, or are breastfeeding
* Clinically significant abnormal physical examination, 12-lead electrocardiogram (ECG) OR cardiac telemetry prior to dosing.
* Significant history or presence of hepatic, renal, cardiovascular, pulmonary, gastrointestinal, hematological, locomotor, immunologic, ophthalmologic, metabolic or oncological disease.
* History or presence of psychiatric or neurologic disease or condition
* History of alcohol or drug abuse
* Any participant who currently uses or has used tobacco or tobacco-containing products for at least one month prior to screening
* Participated in strenuous exercise within 48 hours prior to study start (initial dosing) and/or are unwilling to avoid strenuous exercise at any time throughout the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | Day 1 to Day 21
TS-134 Plasma Pharmacokinetic Profile - Cmax | Cohort 1: Day 1, Day 7, Day 8, Day 14, Cohort 2-3: Day 7, Day 14, Cohort 4-5: Day 9, Day 14, Cohort 6: Day 5, Day 14: predose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, 12h post-dose; Day 1 to Day 14 except above days: predose
  Maximum plasma concentration
TS-134 Plasma Pharmacokinetic Profile - AUC(0-tau) | Cohort 1: Day 1, Day 7, Day 8, Day 14, Cohort 2-3: Day 7, Day 14, Cohort 4-5: Day 9, Day 14, Cohort 6: Day 5, Day 14: predose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, 12h post-dose; Day 1 to Day 14 except above days: predose
  Area under the plasma concentration vs time curve over a dosing interval
TS-134 Plasma Pharmacokinetic Profile - tmax | Cohort 1: Day 1, Day 7, Day 8, Day 14, Cohort 2-3: Day 7, Day 14, Cohort 4-5: Day 9, Day 14, Cohort 6: Day 5, Day 14: predose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, 12h post-dose; Day 1 to Day 14 except above days: predose
  Time to maximum plasma concentration
TS-134 Plasma Pharmacokinetic Profile - t1/2 | Cohort 1: Day 1, Day 7, Day 8, Day 14, Cohort 2-3: Day 7, Day 14, Cohort 4-5: Day 9, Day 14, Cohort 6: Day 5, Day 14: predose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, 12h post-dose; Day 1 to Day 14 except above days: predose
  Apparent terminal elimination half-life
TS-134 Plasma Pharmacokinetic Profile - CL/F | Cohort 1: Day 1, Day 7, Day 8, Day 14, Cohort 2-3: Day 7, Day 14, Cohort 4-5: Day 9, Day 14, Cohort 6: Day 5, Day 14: predose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, 12h post-dose; Day 1 to Day 14 except above days: predose
  Apparent clearance following oral administration
TS-134 Plasma Pharmacokinetic Profile - Vd/F | Cohort 1: Day 1, Day 7, Day 8, Day 14, Cohort 2-3: Day 7, Day 14, Cohort 4-5: Day 9, Day 14, Cohort 6: Day 5, Day 14: predose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, 12h post-dose; Day 1 to Day 14 except above days: predose
  Apparent volumes of distribution following oral administration

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical R&D Inc.
Locations (1):
- PAREXEL - Early Phase Clinical Unit-Los Angeles, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No